CLINICAL TRIAL: NCT02002338
Title: Epidemiological Profile and Comparison Between Different Surgical Techniques for Pterygium Surgery
Brief Title: Different Surgical Techniques for Pterygium Surgery
Status: Completed | Type: Observational
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Sponsor
Other Study IDs: pterygium surgery
Record Dates: First submitted 2013-11-30; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Pterygium
Keywords: pterygium surgery; refractive changes; surgical technique
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pterygium: Patients who were operated of pterygium

SUMMARY:
A study to research the post-operative results according to the chosen surgical technique and evaluate the refractive changes before and after the excision of pterygium.

DETAILED DESCRIPTION:
To analyze the epidemiological profile of patients who were operated of pterygium in Eyes Institute of Goiânia, analyze the post-operative results according to the chosen surgical technique and evaluate the refractive changes before and after the excision of pterygium.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were underwent the pterygium surgery during the period between from February 2013 to August 2013

Exclusion Criteria:

* Patients with mature cataract

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who were underwent pterygium surgery
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Refractive pre-operative | 8 weeks
  Refractive before the excision of pterygium

SECONDARY OUTCOMES:
Refractive post-operative | 8 weeks
  Refractive after the excision of pterygium

OTHER OUTCOMES:
Comparison between different surgical techniques for pterygium surgery | 6 weeks
  To analyze the post-operative results according to the chosen surgical technique and evaluate the refractive changes before and after the excision of pterygium

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R Almeida, MS-V, Study Chair — Instituto de Olhos de Goiania; Larissa S Stival, MD, Study Chair — Instituto de Olhos de Goiania
Locations (1):
- Instituto de Olhos de Goiania, Goiânia, Goiás, Brazil